CLINICAL TRIAL: NCT03898271
Title: Improving Access to Care for Warfighters: Virtual Worlds Technology to Enhance Primary Care Training in Posttraumatic Stress and Motivational Interviewing
Brief Title: PTSD Training for PCPs in a Virtual World
Acronym: VW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Karen Seal, Principal Investigator, San Francisco Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 14-15004
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD; Motivational Interviewing; veterans; military; virtual world; virtual reality; education; training; primary care; mental health
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual World Training (Experimental): Synchronous PTSD training in a virtual world environment
  Interventions: Other: Virtual World
- Web-based Video Training (Active Comparator): Asynchronous web-based PTSD training
  Interventions: Other: Virtual World

INTERVENTIONS:
Other: Virtual World — Participants will complete a synchronous PTSD training in an immersive virtual world environment.

SUMMARY:
The overall goal of this project is improve access to and engagement in quality care for military service personnel and Veterans suffering with posttraumatic stress (PTS). Veterans often present to their primary care providers with symptoms of PTS and related physical problems; however, most primary care providers have not been trained to care for Veterans with PTS or communicate with them in ways that motivate them to engage in care.

In this study instigators propose to design, test and prepare to implement a Virtual World PTS and Motivational Interviewing training for primary care providers by taking the following steps: (1) partner with stakeholders to iteratively design the training which takes full advantage of the affordances of Virtual World technology to enhance training interactivity, effectiveness, and durability, (2) perform a randomized control trial to compare the virtual world training with an online training, and (3) summarize the findings and prepare for implementation and dissemination of the new training by soliciting feedback from primary care providers who participated in the training and from original project stakeholders.

DETAILED DESCRIPTION:
The overall goal of this project is improve access to and engagement in quality care for military service personnel and Veterans suffering with posttraumatic stress (PTS). Veterans who have PTS symptoms after military service are often resistant to referrals to mental health care because of the warrior culture of stoicism coupled with the stigma of seeking mental health care. Also, Veterans living in rural or remote areas may not have access to trained mental health professionals. Thus, Veterans often present to their primary care providers with symptoms of PTS and related physical problems. Unfortunately, most primary care providers have not been trained to care for Veterans with PTS or communicate with them in ways that motivate them to engage in care. This can result in missed opportunities to intervene to prevent what may become chronic mental and physical health problems in the future, which affect not only the warfighter, but also their families, partners and children.

In a prior project funded by the Department of Defense (DoD), study investigators created and tested a web-based training program to teach primary care providers about how to assess for and manage PTS which proved successful in a small pilot study. Nevertheless, primary care providers who participated in the training reported that the training was not interactive and engaging enough and about 30% did not complete it. Moreover, the pilot study did not use gold standard methods to measure study outcomes and because project stakeholders, namely the Veterans Administration (VA) and the DoD, did not participate in the development of the training, investigators were not able to easily implement and disseminate it to primary care clinicians who work in these healthcare systems.

Virtual World technology is a three-dimensional immersive and highly interactive online experience in which users enter virtual environments as self-styled representations of themselves, known as avatars. Virtual Worlds are used in some of the most popular and engaging commercially-available video games. Virtual World technology is also increasingly being used for educational activities, particularly in learning about mental health problems and communication techniques. This is because experiences like mental health symptoms such as re-experiencing or intrusive thoughts (flashbacks) can be simulated, and participants (as avatars) can practice and receive feedback on new communication skills without feeling self-conscious. Learners can also practice motivational interviewing techniques such as using a stylized virtual scale to literally weigh the pros and cons (represented as blocks) of a particular behavior change. These interactive activities afforded by Virtual World technology can be used to make the learning experience far more memorable and enduring.

In this study, investigators propose to design, test and prepare to implement a Virtual World PTS and Motivational Interviewing training by taking the following steps: (1) partner with stakeholders to iteratively design the training so that is responsive to stakeholder needs and takes full advantage of the affordances of Virtual World technology to enhance training interactivity, effectiveness, and durability, (2) add a more robust evaluation component, including a randomized control trial with stronger provider and patient outcomes to achieve more valid results, and (3) summarize findings and prepare for implementation and dissemination of the new training by soliciting feedback from primary care providers who participated in the training and from original project stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* Primary Care Providers (PCPs) currently practicing adult medicine (including licensed internists, family practitioners, nurse practitioners, physician assistants, allied health professionals and trainees working in Primary Care setting)
* English-speaking

Exclusion Criteria:

* Lack of sufficient time to participate in all required training sessions, homework and evaluations.
* Lack of a computer capable of running the Virtual World software
* Retired or retiring during the study period
* Vision or hearing impaired or other disability precluding the use of a computer or telephone*

  * While this is an exclusionary criterion for this trial, prior to broader dissemination, at the conclusion of the study, we will make accommodations in the Virtual World training to make it Section 508-compliant for persons with disabilities.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Motivational Interviewing Treatment Integrity (MITI) Scale | 3 months
  Use standardized patient interviews to observe change in Motivational Interviewing (MI) skills to assess and manage PTSD symptoms and to motivate engagement in care.
PTSD Symptom Assessment and Management Scale | 3 months
  Use standardized patient interviews to observe change in PTSD assessment and management clinical skills.

SECONDARY OUTCOMES:
Evaluation of PTSD Knowledge Questionnaire | 3 months
  Use self-reported measures to observe change in PTSD related knowledge and change in self-reported use of PTSD knowledge after 90 days of no contact.
Self-Efficacy Around PTSD Questionnaire | 3 months
  Use self-reported measures to observe change in PTSD self-efficacy and change in self-reported PTSD self-efficacy after 90 days of no contact.
Provider Satisfaction with Training Questionnaire | 3 months
  Use self-reported measures to compare provider satisfaction with training in the virtual world training vs. the online video training

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco VA Health Care System, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Samuelson KW, Koenig CJ, McCamish N, Choucroun G, Tarasovsky G, Bertenthal D, Seal KH. Web-based PTSD training for primary care providers: a pilot study. Psychol Serv. 2014 May;11(2):153-61. doi: 10.1037/a0034855. Epub 2013 Dec 23. PMID 24364595
- [Derived] Manuel JK, Purcell N, Abadjian L, Cardoos S, Yalch M, Hill C, McCarthy B, Bertenthal D, McGrath S, Seal K. Virtual Worlds Technology to Enhance Training for Primary Care Providers in Assessment and Management of Posttraumatic Stress Disorder Using Motivational Interviewing: Pilot Randomized Controlled Trial. JMIR Med Educ. 2023 Aug 28;9:e42862. doi: 10.2196/42862. PMID 37639299
- See also: Veterans Return Home — http://vetsreturnhome.com/index.html